CLINICAL TRIAL: NCT06746311
Title: Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Characteristics of HT-101 Injection in Healthy Subjects and Patients with Chronic Hepatitis B Virus Infection: a Randomized, Double-blind, Placebo-controlled, Single and Multiple Doses, and Dose Escalation Phase 1 Clinical Study
Brief Title: This is a Phase 1 Study in Which Healthy Volunteers and Participants with Chronic HBV Infection Will Receive HT-101 or Placebo and Will Be Assessed for Safety, Tolerability, Pharmacokinetics (PK), and Antiviral Activity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou HepaThera Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HT-101-101
Record Dates: First submitted 2024-12-09; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part A (Experimental): Single ascending Dose of HT-101 or placebo in Healthy participants subcustaneously.
  Interventions: Drug: HT-101; Drug: Placebo
- Part B (Experimental): Multiple Ascending Dose of HT-101 or placebo in patients with Chronic hepatitis B virus subcustaneously.
  Interventions: Drug: HT-101; Drug: Placebo

INTERVENTIONS:
Drug: HT-101 — Single dose of HT-101 administered subcutaneously.
  Arms: Part A
Drug: HT-101 — Multiple dose of HT-101 administered subcutaneously.
  Arms: Part B
Drug: Placebo — Placebo, containing no active ingredient, administered subcutaneouly

SUMMARY:
Phase 1 Study of HT-101 in Healthy Subjects and Patients With Chronic Hepatitis B The trial consisted of two components. Part A involved a single ascending dose study where healthy participants were administered one dose of HT-101 or placebo subcutaneously (SC). Part B involved a multiple ascending dose study where participants with chronic hepatitis B virus infection were administered two dose of HT-101 or placebo every 4 weeks subcutaneously (SC).

ELIGIBILITY:
Inclusion Criteria: Subjects were eligible for inclusion into the study if they met each of the following criteria:

Part A SAD: Healthy Participant

* Male participants weighed ≥ 50.0 kg, female participants weighed ≥ 45.0 kg;
* Participants who promise having used effective contraception for at least 1 month before screening, and have no plans for pregnancy or donating sperm or eggs, and will voluntarily use effective physical means of contraception (including the partner) during the study and for 3 months after the end of the study;

Part B MAD: Patient with CHB

* Male subjects weighed ≥ 50.0 kg, female subjects weighed ≥ 45.0 kg, with a body mass index (BMI) between 19.0 and 28.0 kg/m^2 (inclusive);
* Chronic HBV infection for >/= 6 months;
* The quantitation level of HBsAg was > 200 IU/mL and < 5000 IU/mL; The quantitation level of HBV DNA < 2×10^4 IU/mL;
* Subjects promised to use effective contraception for at least 1 month before screening, and have no fertility, donate sperm or eggs and voluntarily take highly effective physical contraception (including partners) during the trial and within 3 months after the end of the trial;

Exclusion Criteria:Subjects were excluded from the study if one or more of the following criteria were applicable

* Participants with history of drug allergy or specific allergy;
* Participants who had psychiatric conditions or diseases in cardiovascular, respiratory, endocrine, kidney, liver, digestive tract, skin, immune, blood, nerve and other systems;
* Participants with history of active pathological bleeding, or bleeding tendency;
* Participants with abnormal results of physical examination, vital sign examination, ECG examination, laboratory test in the screening period which were judged as clinically significant by clinicians;
* Participants with significant liver fibrosis or cirrhosis;
* Participants with symptoms or a history of hepatic decompensation;
* Participants with a history or suspected risk of liver cancerr;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | From enrollment to the end of treatment at 24 weeks
  Number of subjects with adverse events (AEs) and serious adverse events (SAEs) assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Clinically significant abnormalities | From enrollment to the end of treatment at 24 weeks
  Number of subjects with clinically significant abnormalities in vital signs, electrocardiogram (ECG), and laboratory parameters graded by CTCAE v5.0.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | From predose 0.5 hours to postdose 48 hours.
  Cmax of HT-101 and its metabolite in plasma. First administration (Healty participants and Patients with CHB): Predose 0.5 hours; Postdose 0.5 hours, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours and 48 hours.
  Second administration (Patients with CHB): Predose 0.5 hours; postdose 0.5 hours, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours and 48 hours.
Time to Reach Maximum Plasma Concentration (Tmax) | From predose 0.5 hours to postdose 48 hours.
  Tmax of HT-101 and its metabolite in plasma. First administration (Healty participants and Patients with CHB): Predose 0.5 hours; Postdose 0.5 hours, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours and 48 hours.
  Second administration (Patients with CHB): Predose 0.5 hours; postdose 0.5 hours, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours and 48 hours.
Area Under the Plasma Concentration Versus Time Curve (AUC) | From predose 0.5 hours to postdose 48 hours.
  AUC of HT-101 and its metabolite from time 0 to last measurable time. First administration (Healty participants and Patients with CHB): Predose 0.5 hours; Postdose 0.5 hours,1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours and 48 hours.
  Second administration (Patients with CHB): Predose 0.5 hours; postdose 0.5 hours,1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours and 48 hours.
Apparent Terminal Elimination Half-life (T1/2) | From predose 0.5 hours to postdose 48 hours.
  T1/2 of HT-101 in plasma. First administration (Healty participants and Patients with CHB): Predose 0.5 hours; Postdose 0.5 hours, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours and 48 hours.
  Second administration (Patients with CHB): Predose 0.5 hours; postdose 0.5 hours, 1hour, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours and 48 hours.
Apparent Plasma Clearance (CL/F) | From predose 0.5 hours to postdose 48 hours.
  CL/F of HT-101 in plasma. First administration (Healty participants and Patients with CHB): Predose 0.5 hours; Postdose 0.5 hours, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours and 48 hours. Second administration (Patients with CHB): Predose 0.5 hours; postdose 0.5 hours, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours and 48 hours.
apparent volume of distribution（Vd/F） | From predose 0.5 hours to postdose 48 hours.
  Vd/F of HT-101. First administration (Healty participants and Patients with CHB): Predose 0.5 hours; Postdose 0.5 hours, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours and 48 hours.
  Second administration (Patients with CHB): Predose 0.5 hours; postdose 0.5 hours, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours and 48 hours.
Maximum Change of Serum HBsAg From Baseline | Up to 24 weeks
  Maximum change of serum HBsAg from Day 1 until 24 weeks post last dose (negative values mean reductions from baseline, positive values mean increased from baseline)
Maximum Change of Serum HBV DNA From Baseline | Up to 24 weeks
  Maximum change of serum HBV DNA from Day 1 until 24 weeks (negative values mean reductions from baseline, positive values mean increased from baseline).
Number of participants with HBeAg Loss | Up to 24 weeks
  For HBeAg-positive Participants: Number of Subjects With HBeAg Loss

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Beijing Ditan Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Nanfang Hospital, Guangzhou, Guangdong
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Yanbian University Hospital, Yanji, Jilin
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No